CLINICAL TRIAL: NCT03360188
Title: Pediatric Multiple Sclerosis in Egypt. A Multi-center Registry of 186 Patients
Brief Title: Pediatric Onset Multiple Sclerosis in Egyptians
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hatem Samir Shehata, professor of Neurology - Cairo University, Cairo University
Other Study IDs: POMS1
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Multiple Sclerosis in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A medical record review of historic and current information on 237 patients attending 5 tertiary referral centers [Kasr Al-Ainy Multiple Sclerosis Research Unit (KAMSU) - Cairo University Hospitals, Abo El Reesh Pediatric Hospital and 3 private centers] in Cairo, Egypt from period between 2011 and December 2015.

Initially, medical records of 251 patients with the first acquired demyelinating events started before age of 18 years were reviewed. Fourteen patients (5.58%) were excluded due to missing data that could not be obtained.

DETAILED DESCRIPTION:
The International Pediatric Multiple Sclerosis Study Group (IPMSSG) criteria were applied on all included patients who were stratified into the following groups: (1) those with 2 or more non-encephalopathic clinical CNS events (NEE) separated by > 30 days and involving > one area of the CNS; (2) one non-encephalopathic episode typical of MS which is associated with MRI findings consistent with 2010 Revised McDonald criteria for dissemination in space and in which a follow up MRI shows at least one new enhancing or non-enhancing lesion consistent with dissemination in time MS criteria; (3) one acute disseminated encephalomyelitis (ADEM) attack followed by a non-encephalopathic clinical event, 3 or more months after symptom onset, that is associated with new MRI lesions fulfilling 2010 Revised McDonald DIS criteria; or (4) a first, single, acute event that does not meet ADEM criteria and whose MRI findings are consistent with the 2010 Revised McDonald criteria for DIS and DIT (applies only to children ≥12 years old).

These criteria were applied retrospectively in patients diagnosed before 2013. Procedures All medical records were analyzed from June 2016 till April 2017 to collect the following data; (1) demographic characteristics; (2) clinical data including age at first symptoms, age at diagnosis, disease course, time to conversion to secondary progressive (SP) course, duration of follow-up, initial and last Expanded Disability Status Scale (EDSS) score, time to (EDSS) score of 4, family history of MS, disease-modifying treatments (DMTs), number of relapses in the first year and the annualized relapse rate (ARR); (3) laboratorial data: oligoclonal bands in the cerebrospinal fluid (CSF) and IgG index; (4) characteristics of the initial magnetic resonance imaging (MRI) of the brain and spinal cord including: typicality of lesions on T2 weighted sequence, presence of brain black holes in T1 weighted sequence, presence of spinal cord T2 lesions, presence of gadolinium (Gd) enhancing lesions, distribution of brain lesions (supratentorial and/or infratentorial).

Data quality. To ensure high-quality data, the accuracy and completeness were systemically assessed. The medical records, administrative data, laboratory and diagnostic tests reports were screened independently by 2 authors (NS and AE) and relevant data was extracted to a standard electronic form according to KAMSU registry. An assigned coordinator from each center was requested to facilitate data collection from site-specific records; an audit site-specific data abstractor was continuously monitoring the records. Data accuracy was checked by separate investigators (MA, HS, AH) who reviewed the electronic forms for resemblance. Scheduled monthly meetings between abstractors were held to resolve any data conflicts. In case of incomplete documentation or unclear information, verification was done by the on-site data coordinator either by phone or during a face-to-face interview with the patients or caregivers during routine follow up or unscheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* All included patients had the onset of the first symptoms before the age of 18 years; and they were further classified into (1) below 12 years old or early-onset pediatric multiple sclerosis (EOPMS), and (2) ≥12 years old or late-onset pediatric MS (LOPMS) according to The International Pediatric Multiple Sclerosis Study Group (IPMSSG) criteria

Exclusion Criteria:

* MS mimics

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 237 patients were finally analyzed in the current study, 64.56% (153) were females and 35.44% (84) were males. At time of data collection; MS was diagnosed in 186 patients (78.48%); and the diagnosis of 10 patients (4.22%) were not yet settled. We identified 47/186 patients (25.27%) with EOPMS. Positive family history of MS [at least one first and/or second degree relatives] was reported in 15/186 patients (8.06%). The median (IQR) time between the first manifestation and confirmation of the diagnosis was 6 months (3 - 9) months.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
time to EDSS 4 | up to 150 months
  The time to EDSS 4 from symptoms onset in relation to initiation of Disease Modified Therapies (before/after 1 year of symptoms onset)

IPD SHARING:
Plan to Share IPD: No